CLINICAL TRIAL: NCT01779986
Title: Comparison of the Evaluation of CAD by CT AngioScan and Coronary Angiogram in Patient as Part of Preoperative Evaluation in Ascending Aorta Replacement Surgery Patients.
Brief Title: Comparison of the Evaluation of CAD by CT AngioScan and Coronary Angiogram
Acronym: CTAS-MCAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: CTAS-MCAS UdeS 12-073
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of CT Coronary Angioscan (CT-AS) is gaining popularity, but its exact value as evaluation of CAD requires confirmation. We intend to compare the results of CT-AS and convention coronary angiogram results in patients who are scheduled for an ascending aorta aneurysm reparation surgery. These examens are standard of care before this surgery, so there is no additional danger or disadvantage for the patient. We hope to confirm that CT-AS is a reliable screening test for CAD in patient undergoing heart surgery for other reason than CAD.

ELIGIBILITY:
Inclusion Criteria:

* Ascending aorta aneurysm waiting for surgical correction
* Willing to participate
* Needing a Coronary angiogram and a CT-AS for medical reasons

Exclusion Criteria:

* Refuse to participate
* Allergy to contrast material
* Incomplete results or having one of the test done in another hospital
* Arrythmia
* More than 6 months between the two exams

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ascending aorta aneurysm undergoing preoperative evaluation of CAD by CT-Angioscan and Coronary angiogramm before surgical reparation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Presence of CAD | less than 6 monthes between two tests
  The CAD seen on CT-AS as compared to the results of the gold-standard test of coronary angiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gahide, MD PHD, Principal Investigator — Université de Sherbrooke
Locations (1):
- CHUS Fleurimont, Sherbrooke, Quebec, Canada